CLINICAL TRIAL: NCT03708536
Title: Bevacizumab Plus Capecitabin vs S-1 as Maintenance Treatment Following First-line Chemotherapy in the Patients With Advanced Colorectal Adenocarcinoma. A Phase 3 Randomised Controlled Trial
Brief Title: Bevacizumab Plus Capecitabin vs S-1 as Maintenance Treatment Following First-line Chemotherapy in the Patients With Advanced Colorectal Adenocarcinoma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: There are no fund to support
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNF 012
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2018-10

CONDITIONS: Colorectal Adenocarcinoma
Keywords: bevacizumab; s-1; capecitabin; maintenance
MeSH Terms: interventions — S 1 (combination); Bevacizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bevacizumab plus s-1 (Experimental)
  Interventions: Drug: S-1
- bevacizumab plus capecitabin (Active Comparator)
  Interventions: Drug: Bevacizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: S-1 — S-1 is administered orally on days 1 to 14 of a 21-day cycle. Patients are assigned on the basis of body surface area (BSA) to receive one of the following oral doses twice daily: 40 mg (BSA <1.25m2), 50 mg (BSA >1.25 to <1.50 m2), or 60 mg (BSA >1.50 m2).
  Arms: bevacizumab plus s-1
Drug: Bevacizumab — Bevacizumab (7.5 mg/kg) is administered by intravenous infusion over the course of 30 to 90 min on day 1 of each 3-week cycle.
  Arms: bevacizumab plus capecitabin
Drug: Capecitabine — Capecitabine 2000mg/m2/d is administered orally on days 1 to 14 of a 21-day cycle.
  Arms: bevacizumab plus capecitabin

SUMMARY:
Bevacizumab plus capecitabin is a standard maintenance treatment following first-line chemotherapy in the patients with advanced colorectal adenocarcinoma. However, hand-foot syndrome induced by capecitabin will bother the patient to decrease the quality of life. S-1, an alternative of fluoropyrimidine, was proved non-inferior efficacy with lower hand-foot syndrome as first-line chemotherapy in advanced colorectal adenocarcinoma in the studies. The investigators are going to test the efficacy and safety of bevacizumab plus S-1 as maintenance treatment compared with bevacizumab plus capecitabin in colorectal adenocarcinoma

ELIGIBILITY:
Criteria

Before the start of induction therapy:

Inclusion Criteria:

Histological proof of colorectal cancer (in case of a single metastasis, histological or cytological proof of this lesion should be obtained); Distant metastases (patients with only local recurrence are not eligible); Unidimensionally measurable disease (> 1 cm on spiral CT scan or > 2 cm on chest X-ray; liver ultrasound is not allowed). Serum CEA may not be used as a parameter for disease evaluation; In case of previous radiotherapy, at least one measurable lesion should be located outside the irradiated field.

Ongoing or planned first line treatment with 6 cycles of Xeloda, Eloxatin, and Avastin.

Exclusion criteria Prior adjuvant treatment for stage II/III colorectal cancer ending within 6 months before the start of induction treatment Any prior adjuvant treatment after resection of distant metastases Previous systemic treatment for advanced disease

At randomisation:

Inclusion criteria:

WHO performance status 0-1 (Karnofsky PS > 70%); Disease evaluation with proven SD, PR or CR according to RECIST after 6 cycles of MTD chemotherapy performed in week 3-4 of the 6th cycle induction therapy, and randomisation performed in week 3-5 of the 6th cycle (see time table); Laboratory values obtained ≤ 2 weeks prior to randomisation: adequate bone marrow function (Hb > 6.0 mmol/L, absolute neutrophil count > 1.5 x 109/L, platelets > 100 x 109/L), renal function (serum creatinine ≤ 1.5x ULN and creatinine clearance, Cockroft formula, > 30 ml/min), liver function (serum bilirubin ≤ 2 x ULN, serum transaminases ≤ 3 x ULN without presence of liver metastases or ≤ 5x ULN with presence of liver metastases); Life expectancy > 12 weeks; Age >= 18 yrs; Negative pregnancy test in women with childbearing potential; Expected adequacy of follow-up; Institutional Review Board approval; Written informed consent Exclusion criteria History or clinical signs/symptoms of CNS metastases; History of a second malignancy ≤ 5 years with the exception of adequately treated carcinoma of cervix or basal/squamous cell carcinoma of skin; Previous intolerance of XelodaR, EloxatinR, and/or AvastinR for which any of these drugs have been permanently discontinued; patients with previous dose reductions or delays are eligible; patients with grade 2 neurotoxicity after the 6th cycle are eligible, and retreatment with EloxatinR after PFS1 should depend on the grade of neurotoxicity at that moment; Known dihydropyrimidine dehydrogenase (DPD) deficiency; (Planned) radical resection of all metastatic disease; Uncontrolled hypertension, i.e. consistently > 150/100 mmHg; Use of more than 3 antihypertensive drugs; Significant cardiovascular disease < 1 yr before randomisation (symptomatic congestive heart failure, myocardial ischemia or infarction, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, arterial thrombosis, cerebrovascular event, pulmonary embolism); Any of these significant cardiovascular events during previous fluoropyrimidine therapy; Chronic active infection; Any other concurrent severe or uncontrolled disease preventing the safe administration of study drugs; Any impairment of gastrointestinal function or -disease that may significantly impair the absorption of oral drugs (i.e. uncontrolled nausea, vomiting, diarrhoea (defined as >CTC grade 2), malabsorption syndrome, bowel obstruction, or inability to swallow tablets); Concomitant treatments: concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation; concurrent treatment with any other anti-cancer therapy; full-dose anticoagulation (is allowed if started during induction therapy); Continuous use of immunosuppressive agents (except the use of corticosteroids as anti-emetic prophylaxis/treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment to progression of disease. Estimated about 6 months.
  The length of time from enrollment until the time of progression of disease

SECONDARY OUTCOMES:
Overall survival | From enrollment to death of patients. Estimated about 1 year.
  The length of time from enrollment until the time of death

OTHER OUTCOMES:
Toxicity | From enrollment to 3 months after treatment
  According to NCI CTCAE 4.03 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Rongbo Lin, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No